CLINICAL TRIAL: NCT07375147
Title: Outcomes of Transanal Versus Transvaginal Rectal Resection for Anterior Rectocele: A Randomized Controlled Trial
Brief Title: Transanal vs Transvaginal Rectal Resection for Anterior Rectocele
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abdelaal, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD-133-2025
Record Dates: First submitted 2026-01-12; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-06

CONDITIONS: Rectocele; Female
Keywords: Rectocele; Obstructed defecation; Stapled Transanal Rectal Resection; Stapled Transvaginal Rectal Resection
MeSH Terms: conditions — Rectocele

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stapled Transanal Rectal Resection (Active Comparator): Patients in this group will be conducted to Stapled Transanal rectal resection for the anterior rectocele
  Interventions: Procedure: Stapled Transanal Rectal Resection
- Stapled Transvaginal Rectal Resection (Experimental): patients in this group will be conducted to stapled transvaginal rectal resection for the anterior rectocele
  Interventions: Procedure: Stapled Transvaginal Rectal Resection

INTERVENTIONS:
Procedure: Stapled Transanal Rectal Resection — Patients were placed in the lithotomy position. Using the trans-anal approach, rectocele was done using PPH circular staplers. A circular anal dilator (CAD) was inserted into the anus and sutured into position. Three full-thickness prolene 2/0 sutures were positioned at the anterior, left anterior lateral, and right anterior lateral locations, approximately 4 cm above the dentate line. At the posterior aspect, a tongue depressor was placed into the CAD groove to protect the posterior rectal wall. After insertion of the Procedure for Prolapse and Hemorrhoids stapler (PPH stapler) into the rectum with its head open past the proximal suture, PPH stapler was progressively closed. Per vaginal examination was done To make sure the stapler did not include the vagina. The stapler was then fired to complete the anterior rectal resection.
  Arms: Stapled Transanal Rectal Resection
Procedure: Stapled Transvaginal Rectal Resection — The patient in the lithotomy position. Anal dilatation was performed. A transverse incision was made in the mucocutaneous border of the vaginal introitus; the posterior vaginal wall was dissected and separated from the anterior rectal wall up to the posterior fornix. Dissection was extended laterally to the maximum length of the rectocele. Two Babcock clamps were applied longitudinally to the rectocele, and the stapler was fired to divide the rectocele. Partial thickness stitches were applied over the staple line using vicryl 2/0 suture to reinforce the staple line.
  Arms: Stapled Transvaginal Rectal Resection

SUMMARY:
Female patients presenting with obstructed defecation syndrome due to anterior rectocele will be screened according to inclusion and exclusion criteria. Eligible patients will undergo clinical assessment and appropriate investigations including defecography. After informed consent, patients will be randomized into two groups: Stapled Transanal rectal resection or Stapled Transvaginal rectal resection. Improvement in obstructed defecation symptoms and postoperative complications will be compared between the two groups.

DETAILED DESCRIPTION:
This is a randomized controlled trial aims to compare the clinical outcomes of Stapled Transanal versus Stapled Transvaginal rectal resection in female patients with obstructed defecation syndrome (ODS) caused by anterior rectocele.

Female patients presenting to the outpatient colorectal clinic with symptoms of obstructed defecation syndrome will be screened for eligibility according to predefined inclusion and exclusion criteria. All eligible patients will receive a detailed explanation of the study objectives, procedures, potential benefits, and risks. Written informed consent will be obtained prior to enrollment.

A comprehensive preoperative evaluation will be performed for all participants, including detailed medical history, physical and anorectal examination, and appropriate investigations including defecography to confirm the diagnosis and assess the severity of rectocele.

Enrolled patients will be randomly assigned in a 1:1 ratio into one of two intervention groups. Group A will undergo stapled Transanal rectal resection, while Group B will undergo stapled transvaginal rectal resection. All surgical procedures will be performed by experienced colorectal surgeons.

Primary outcome measures will include improvement in obstructed defecation symptoms as assessed by Cleveland Clinic Constipation (CCC) score. Secondary outcomes will include length of hospital stay, operative time, postoperative pain score, postoperative continence state, Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients complaining of obstructed defecation syndrome with anterior rectocele ≥ 3 cm on straining with failure of conservative management.

Exclusion Criteria:

* Patients with Slow-transit constipation
* Patients with rectocele of < 3 cm on straining
* Patients with complete external rectal prolapse
* Evidence of colorectal carcinoma or Inflammatory bowel disease ( IBD)
* Previous rectal surgeries
* Inability for lifestyle change postoperatively
* Previous surgeries for anterior rectocele

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-06-14 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in obstructed defecation symptoms in both groups using Cleveland Clinic Constipation (CCC) score | Up to 6 months postoperatively
  Compare Improvement in obstructed defecation symptoms in both groups using Cleveland Clinic Constipation (CCC) score. CCC score ranges from 0 to 30. Higher scores indicate a worse outcome (more severe obstructed defecation symptoms )

SECONDARY OUTCOMES:
Operative time | During surgery
  Compare time of operation between both procedure
Hospitalization period | From date of hospital admission until date of hospital discharge, assessed up to 10 days after surgery
  Compare how many days patients stay in hospital in both groups
surgical site infection | Up to 6 months postoperatively
  compare surgical site infection in both groups
Time for wound Healing | Up to 6 months postoperatively
  Time for wound Healing in both groups
Postoperative bleeding | Up to 6 months postoperatively
  Compare Postoperative bleeding in both groups
Postoperative fecal incontinence | Up to 6 months postoperatively
  Compare post postoperative fecal incontinence in both groups
Postoperative urine retention | Within 48 hours postoperatively
  Compare postoperative urine retention in both groups
Pain intensity | At day 1 and day 7 postoperatively
  Compare Pain intensity measured using Visual Analogue Scale between both groups (Visual Analogue Scale for Pain: ranges from 0 to 10 . Higher scores indicate a worse outcome {greater pain intensity})
Sexual Function in both groups | Up to 6 months postoperatively
  Compare sexual function in both groups using Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ- 12). PISQ-12 score ranges from 0 to 48. Higher scores indicate better sexual function
Postoperative anal stenosis in both groups | Up to 6 months postoperatively
  Postoperative anal stenosis will be assessed by digital rectal examination and graded clinically as follows:
  * Mild: anal canal admits a well lubricated index finger.
  * Moderate: Forceful dilatation required to admit a well lubricated index finger.
  * Severe: Little finger cannot be admitted without forceful dilatation
Postoperative rectovaginal fistula in both groups | Up to 6 months postoperatively
  Postoperative rectovaginal fistula will be assessed using the following methods:
  * History: Passage of flatus or stool from the vagina.
  * Clinical examination: Digital rectal examination and per vaginal examination to detect induration or fistula opening.
  * MRI of the pelvis: Performed if fistula is suspected based on history or clinical examination to confirm the diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Tamer, lecteurer, Study Director — Cairo University
Locations (1):
- Faculty of medicine, Cairo University, Cairo, Al-Manial, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this is a small surgical trial with a limited number of participants, and sharing raw data could lead to identification of participants